CLINICAL TRIAL: NCT05375526
Title: Magtrace® as Tracer for Sentinel Lymph Node Detection in Early Stage Epithelial Ovarian Cancer: a Pilot Study
Brief Title: Magtrial: Magtrace® as Tracer for Sentinel Lymph Node Detection in Early Stage Epithelial Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL75863.068.21
Record Dates: First submitted 2022-05-05; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer; Lymph Node Metastasis
Keywords: Sentinel lymph node
MeSH Terms: conditions — Ovarian Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary staging laparotomy for suspicion of early stage EOC (Experimental): In case of a primary staging laparotomy the diagnosis of malignancy is based on a frozen section of the resected adnexa, followed by the sentinel node technique during the same procedure.
  Interventions: Device: Magtrace
- Secondary staging laparotomy for EOC (Experimental): On the other hand, in some cases early stage EOC is only diagnosed after the primary surgery, when the surgeon resects the ovary with the suspicion of benign disease. If the adnexa are already removed before the diagnosis of malignancy, a secondary staging laparotomy is required and, in this case, a single step approach for SLN is not feasible.
  Interventions: Device: Magtrace

INTERVENTIONS:
Device: Magtrace — In the proper ovarian ligament (or its remnants), close to the ovary and just below the peritoneum Magtrace® will be injected via a 12 Gauge (2mm) needle. This injection will be followed by an injection of 20 MBq 99mTc via the same 12 Gauge (2mm) needle.
  If a hysterectomy has been conducted, this step can be omitted. In the infundibulopelvic ligament (suspensory ligament of the ovary), close to the ovary and just below the peritoneum Magtrace® will be injected via a 12 Gauge (2mm) needle. This injection will be followed by an injection of 20 MBq 99mTc via the same 12 Gauge (2mm) needle.

SUMMARY:
Epithelial ovarian cancer (EOC) remains the tumour with the most unfavourable prognosis within the field of gynaecological oncology. The incidence of ovarian cancer in the Netherlands in 2008 was 14.5 per 100.000, with 12.3 deaths per 100.000. In the US in 2007 the incidence was 13.0 per 100.000 and there were 8.2 deaths per 100.000. The high mortality rate is partially due to the fact that approximately 75% of patients is diagnosed with advanced stage EOC. The remaining 25% of patients are diagnosed in an early stage, which require a complete surgical staging procedure including pelvic and para-aortic lymphadenectomy. Although this lymphadenectomy is standard-of-care, it leads to significant morbidity in these patients. Mainly direct postoperative complications such as infection, repeat surgery and early death have been reported. Also, long-term complications such as lymph cysts or lymphedema have been described.

A potential method to reduce this morbidity and mortality, as already been described in other cancers such as breast cancer and vulvar cancer, is utilizing a sentinel lymph node (SLN) technique. By identifying and resecting the SLN, the patient is potentially spared form lymphadenectomy.

DETAILED DESCRIPTION:
Background EOC can metastasize through three different pathways: intraperitoneal (in the abdominal cavity), lymphogenous or haematogenous [5,6]. Concerning the lymphogenous spread, it is clear that lymphatic spread of EOC occurs mainly to the para-aortic lymph nodes. It is theorized that the tumour cells follow the lymph vessels that accompany the ovarian vessels in the infundibulopelvic ligament up to the upper para-aortic region and renal vein. Additionally, pelvic lymph node metastases are also frequently found. These tumour cells probably follow a different route, migrating via the para-uterine vessels in the broad ligament towards the uterine vessels and further on to the iliac vessels and lymph nodes. In some case reports, isolated inguinal node metastases are also described. The exact mechanism of this route of metastasis is still unclear, but the metastatic cells might follow the course of the round ligament towards the inguinal lymph nodes or follow the iliac vessels towards the femoral vessels.

According to the International Federation of Gynaecology and Obstetrics (FIGO), EOC with lymph node metastases is classified as FIGO stage IIIA1. This significant upstaging is reflected in the need for adjuvant treatment. While patients with cancer confined to the ovaries (FIGO stage I) do not require adjuvant chemotherapy, patients with EOC FIGO stage III require additional treatment. Therefore, the detection of lymph node metastases is of utmost importance in perceived early stage disease.

In case of a clinical early stage ovarian cancer, standard-of-care is a staging laparotomy including bilateral pelvic and para-aortal lymphadenectomy. There is 14% (range 6.1-29.6%) chance of finding lymph node metastases . The incidence is higher in the grade 3 tumours (20.0%) and the serous histological subtype (23.3%). Whereas in grade 1 and mucinous tumours this is respectively 4.0% and 2.6%. By removing a greater number of lymph nodes, the detection rate for metastases rises . Although complete pelvic and para-aortic lymphadenectomy is standard-of-care, radical lymphadenectomy has been associated with serious morbidity and this is a major reason for the difference in the extent of lymph node dissection between centres.

By resecting only the SLN, significant reduction of morbidity and mortality can be obtained in comparison with the standard-of-care. SLN surgery is based on the concept that, if the SLN has no malignant cells, the likelihood that other lymph nodes are affected is reduces to almost non-existent. This means that, at least theoretically, a radical lymphadenectomy could be omitted and thus the associated morbidity and potential mortality. The SLN technique has been proven to be effective in other cancers such as breast cancer and malignant melanoma. In the gynaecological field it has been shown to be effective in vulvar cancer. Several SLN studies have been conducted in patients with ovarian cancer with promising results, as summarized in Table 1.

Rationale As stated, the goal of utilizing SLN in early-stage EOC surgery is to reduce patient morbidity while obtaining optimal oncological outcomes. By resecting only the SLN, the patients would be spared from radical lymphadenectomy, reducing short and long-term complications.

As summarized in Table 1, most studies utilize 99mTc and blue dye to visualize the SLN. Although detection rates are good with these techniques, they have major disadvantages. 99mTC is an isotope, as such it exposed the patient to an irradiation dose. Although total dosage is limited, eliminating isotopes in surgery would reduce the potential harm for the patient and the medical staff during surgery. Furthermore, the process to produce and administer 99mTC is a costly and resource-intensive procedure, requiring the cooperation of nuclear medicine, radio-pharmacy and logistics. As such, reducing the need for 99mTc would benefit the patient, medical staff and the healthcare system in general by reducing costs. Blue dye such as Patent Blue is often used for the detection of SLN. However, it also has major disadvantages. Firstly, it potentially occludes the entire operation field because of dissemination of the dye further than the SLN. Without optimal visualisation of the anatomy, the surgeon can expect more difficult dissection. Secondary, blue dye can cause a severe allergic reaction, leading to anaphylactic shock in up to 2% of patients.

Magtrace® is a brownish ferromagnetic substance capable of identifying the SLN. This novel technique has already been extensively researched in breast cancer and proven to be non-inferior to 99mTc with blue dye. These promising results led to licensing in the European Union. In this trial, the investigators wish to examine the potential of this technique in EOC, eliminating the disadvantages of 99mTc and blue dye. However, this is still a pilot study with unknown efficacy in EOC. Therefore, in order to minimize potential harm to the patient, 99mTc will be co administrated. This has been deliberately chosen due to the extensive literature concerning this sentinel mapping technique (see Table 1). If the efficacy of Magtrace would prove successful, the ultimate goal is to omit 99mTc in further studies and use Magtrace® only to identify the SLN.

In this pilot study, researchers will include two study arms. One in primary staging laparotomy, the other one in secondary staging laparotomy. The rationale of these two arms is based on the clinical practice, were surgeons not always suspect malignancy before resection of the adnexa. In case of a primary staging laparotomy the diagnosis of malignancy is based on a frozen section of the resected adnexa, followed by the sentinel node technique during the same procedure. On the other hand, in some cases early stage EOC is only diagnosed after the primary surgery, when the surgeon resects the ovary with the suspicion of benign disease. If the adnexa are already removed before the diagnosis of malignancy, a secondary staging laparotomy is required and, in this case, a single step approach for SLN is not feasible. The design of two study arms in this pilot study allows to compare the efficacy of Magtrace in native tissue (primary staging laparotomy) with tissue afflicted by previous surgery (secondary staging laparotomy).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a high suspicion of an early stage malignant EOC planned for exploratory laparotomy.
* Patients with a confirmed early stage malignant EOC where a secondary staging laparotomy will be performed.
* Age between 18 and 85 years.

Exclusion Criteria:

* Secondary staging laparotomy for stage I expansile type mucinous adenocarcinoma.

  * Patients with suspicion of positive lymph nodes in the inguinal, pelvic, para-aortal or other lymph regions (either clinically or radiographically).
  * Patients with suspicion of metastasis (either clinically or radiographically).
  * Patients with previous ovarian surgery.
  * Patients with previous vascular surgery of the aorta, inferior vena cava, and/or iliac vessels.
  * Patients with previous lymphadenectomy of lymph node sampling in the iliac or para-aortal region.
  * Patients with history of a malignant lymphoma.
  * Patients with history of a malignant tumour in the abdominal cavity other than EOC
  * Patients who are pregnant or lactating.
  * Patients with an allergy for human albumin.
  * Patients have had preoperative radiation therapy to the pelvis.
  * Patients with an iron overload disease.
  * Patients with intolerance or hypersensitivity to iron or dextran compounds or to Magtrace®.
  * Patients with a metal implant close to the expected sentinel lymph node location.
  * Patients who are deprived of liberty or under guardianship.
  * Patients not able to follow and understand the procedures of the study due to mental state or other reasons.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer is a female only disease
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
To assess the use of Magtrace® as a tracer in SLN sampling in early stage EOC | 2 years
  Can sentinel lymph nodes be found using magtrace this means a positive signal. The patient will have a interpatient control using radio active technetium. Outcome will be reported as: Magtrace found sentinel lymph node: yes or no

SECONDARY OUTCOMES:
Comparison of detection rate between MagTrace® and 99mTc | 2 years
  Between 1 primary staging laparotomy and 2 in secondary staging laparotomy
Detection of potential adverse effects of MagTrace® and 99mTc | 2 years
Relationship between the observed SLN and the actual number of pathological lymphnodes | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR